CLINICAL TRIAL: NCT02816762
Title: Effect of Continuous Positive Airway Pressure on Albuminuria in Patients With Diabetic Nephropathy and Obstructive Sleep Apnea
Brief Title: CPAP Effect on Albuminuria in Patients With Diabetic Nephropathy and Obstructive Sleep Apnea
Acronym: DIANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP
Record Dates: First submitted 2016-05-31; First posted 2016-06-29 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Nephropathy; Sleep Apnea
Keywords: CPAP; Sleep apnea; Diabetes; Nephropathy; Albuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Sleep Apnea Syndromes; Diabetes Mellitus; Kidney Diseases; Albuminuria | interventions — Continuous Positive Airway Pressure; Drug Therapy; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP treatment (Experimental): Diet and conventional pharmacological treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists or anti-aldosterone agents plus continuous positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure; Drug: Pharmacological treatment; Other: Diet
- Control treatment (Active Comparator): Diet and conventional pharmacological treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists or anti-aldosterone agents.
  Interventions: Drug: Pharmacological treatment; Other: Diet

INTERVENTIONS:
Device: Continuous positive airway pressure — Nocturnal continuous positive airway pressure by a nasal mask. CPAP pressure will be automatically titrated using a AutoSet device (ResMed).
  Arms: CPAP treatment
Drug: Pharmacological treatment — Conventional pharmacological treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists or anti-aldosterone agents.
  Other Names: Conventional pharmacological treatment
Other: Diet — Conventional anti-diabetic diet recommendations

SUMMARY:
Objectives: Main objective: To assess the effect of 12 months of CPAP treatment added to conventional drug treatment on the albuminuria in patients with diabetic nephropathy and obstructive sleep apnea (OSA). Secondary objectives: To evaluate the effect of CPAP treatment on the estimated glomerular filtration rate of patients with diabetic nephropathy and OSA; determine the additional longterm CPAP effect on glycemic control, insulin resistance, lipid profile, health-related quality of life and biomarkers of cardiac function, inflammation, oxidative stress, sympathetic tone and appetite-regulating hormones in patients with diabetic nephropathy and OSA; and to identify the subgroup of patients with diabetic nephropathy and OSA in which 12 months of treatment with CPAP achieve a more pronounced reduction in albuminuria.

Methodology: Randomized, multicenter, non-blinded, parallel groups, conventional treatment-controlled trial of 12 months of duration.

Subjects will randomize to conventional dietary and pharmacological treatment or conventional dietary and pharmacological treatment plus continuous positive airway pressure (CPAP). Study subjects: Subjects 18 to 80 years with overweight or obesity and a clinical diagnosis of diabetic nephropathy, increased urinary albumin/creatinine ratio of 30 mg/g and an estimated glomerular filtration rate >20 ml/min/1.73 m2, and treatment with stable doses of angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers (ARBs) or anti-aldosterone drugs in the last four weeks. Efficacy variables:

urinary albumin/creatinine ratio and estimated glomerular filtration rate; glycosylated hemoglobin (HbA1c); fasting glucose and insulin; homeostatic model assessment (HOMA) and QUICKI indices; total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides; Troponin I, proBNP, homocysteine and high-sensitivity C-reactive protein; systemic biomarkers (inflammation [IL-6, IL-8 and tumor necrosis factor-α], oxidative stress [8-isoprostane], endothelial damage [endothelin, VCAM-1 and ICAM-1], sympathetic activity [neuropeptide Y] and appetite-regulating hormones [leptin and adiponectin]) and clinical questionnaires: short form (SF)-12, EuroQoL and iPAQ.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 80 years old
* Overweight or obesity (BMI ≥25 kg/m2)
* Previous diagnosis of type 2 diabetes, fulfilling at least one of the following criteria: 1) current treatment with oral antidiabetic drugs and/or insulin; 2) a fasting glucose value above 126 mg/dl on at least 2 occasions; 3) blood glucose level at 2 hours after an oral glucose tolerance test is equal to or more than 200 mg/dl; or 4) a glycated hemoglobin (HbA1c) level > 6.5 %
* Clinical diagnosis of diabetic nephropathy, with a urinary albumin/creatinine ratio >30 mg/g and an estimated glomerular filtration rate more than 20 ml/min per 1.73 m2.
* Treatment with stable doses of angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers or anti-aldosterone agents in the last four weeks.

Exclusion Criteria:

* Non diabetic nephropathy (confirmed by biopsy).
* Dialysis for acute renal failure within the 6 previous months.
* Evidence in the clinic history of relevant bilateral stenosis of renal artery (> 75%)
* Urinary albumin/creatinine ratio higher than 3000 mg/g, at the baseline visit.
* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mm Hg at the baseline visit.
* Stroke, transient ischemic attack, acute coronary syndrome, or hospitalization for heart failure worsening, within the previous 30 days.
* Professional drivers, risk profession or respiratory failure.
* Severe daytime sleepiness (Epworth sleepiness scale >18)
* Concomitant treatment with high doses of acetylsalicylic acid (> 500 mg/day) or continuous treatment with non-steroidal anti-inflammatory drugs
* Previous treatment with CPAP
* Participation in another clinical trial within the 30 days prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change form baseline in albuminuria levels | 12 months
  To compare the change in albuminuria levels between the patients allocated to CPAP group and the control group

SECONDARY OUTCOMES:
Change from baseline in glycated hemoglobin levels | 12 months
  To compare the change in glycated hemoglobin levels between the patients allocated to CPAP group and the control group
Change form baseline in HOMA index | 12 months
  To compare the change in HOMA index between the patients allocated to CPAP group and the control group
Change form baseline in QUICKI index | 12 months
  To compare the change in QUICKI index between the patients allocated to CPAP group and the control group
Change from baseline in cholesterol levels | 12 months
  To compare the change in the levels of total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides between the patients allocated to CPAP group and the control group
Change from baseline in the levels of C-reactive protein | 12 months
  To compare the change in the levels of C-reactive protein between the patients allocated to CPAP group and the control group
Change from baseline in the health-related quality of life assessed by the SF-12 questionnaire | 12 months
  To compare the change in the total score and the domains of the questionnaire SF-12 between the CPAP group and the control group
Change from baseline in the health-related quality of life assessed by the EuroQoL questionnaire | 12 months
  To compare the change in the total score and the domains of the questionnaire EuroQoL between the CPAP group and the control group
Change from baseline in the daily physical activity of patients with diabetic nephropathy and OSA | 12 months
  To compare the change in the total score of the International Physical Activity Questionnaire (iPAQ) between the CPAP group and the control group
Change form baseline in the plasmatic levels of biomarkers of inflammation | 12 months
  To compare the change in the plasmatic levels of interleukin (IL)-1beta, IL-6, IL-8 and tumor necrosis factor-alpha between the CPAP group and the control group
Change form baseline in the plasmatic levels of 8-isoprostane | 12 months
  To compare the change in the plasmatic levels of 8-isoprostane between the CPAP group and the control group
Change form baseline in the plasmatic levels of endothelin | 12 months
  To compare the change in the plasmatic levels of endothelin, intercellular adhesion molecule-1 (ICAM-1) and vascular cell adhesion molecule-1 (VCAM-1) between the CPAP group and the control group
Change form baseline in the plasmatic levels of appetite-regulating hormones | 12 months
  To compare the change in the plasmatic levels of leptin and adiponectin between the CPAP group and the control group
To identify the CPAP-responder subgroup of OSA patients with diabetic nephropathy | 12 months
  To identify the subgroup of OSA patients with diabetic nephropathy in those the CPAP treatment achieve an albuminuria reduction >20% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Study Chair — Hospital Universitario La Paz, IdiPAZ
Locations (6):
- Spain (6):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario General de Guadalajara, Guadalajara
  - Hosptial Universitario La Paz, IdiPAZ, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zamarron E, Jaureguizar A, Garcia-Sanchez A, Diaz-Cambriles T, Alonso-Fernandez A, Lores V, Mediano O, Troncoso-Acevedo F, Cabello-Pelegrin S, Morales-Ruiz E, Ramirez-Prieto MT, Valiente-Diaz MI, Gomez-Garcia T, Casitas R, Martinez-Ceron E, Galera R, Cubillos-Zapata C, Garcia-Rio F. Continuous Positive Airway Pressure Effect on Albuminuria Progression in Patients with Obstructive Sleep Apnea and Diabetic Kidney Disease: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2023 Mar 15;207(6):757-767. doi: 10.1164/rccm.202206-1091OC. PMID 36342964